CLINICAL TRIAL: NCT06691009
Title: Effectiveness of Pleurodesis by Pleural Abrasion Using Medical Thoracoscopy Versus Bleomycin Via Pleural Catheter in Patients With Malignant Pleural Effusion
Brief Title: Pleural Bleomycin vs Mechanical Abrasion in Malignant Pleural Effusion
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Mahmoud Mohammed Eltayeb, Assistant lecturer of chest diseases, Assiut University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: Interventions for MPE
Record Dates: First submitted 2024-08-17; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-10

CONDITIONS: Malignant Pleural Effusion
MeSH Terms: conditions — Pleural Effusion, Malignant

STUDY DESIGN:
Intervention Model Description: Random assignment of intervention will be done after subjects have been assessed for eligibility and recruited and after final diagnosis. This will be done by crossover method 1:1. Patients with ODD number will be included in group 1, and patients with even number will be included in group 2.
Who Masked: Participant, Outcomes Assessor
Masking Description: There will be an outcome assessor who do not know which group recieved which treatment. Also, the participants will not know to which group they will be included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Mechanical pleurodesis) (Experimental): Pleural abrasions will be done by scrubbing the parietal and visceral pleura until a uniform aspect of bloody pleura by a piece of gauze attached to the end of a holding forceps, and intercostal tube will then placed and monitoring of lung expansion will be done through serial CXR and chest ultrasound follow up and when the lung is fully expanded the tube will be clamped for two hours and follow up CXR will be done for follow up and then the tube removed.
  Interventions: Procedure: Group 1 (mechanical pleurodesis)
- Group 2 (Chemical pleurodesis by bleomycin) (Experimental): Those Patients will have indwelling pleural catheter through which pleural fluid will be drained until dryness and then pleurodesis will be done by 60 mg bleomycin dissolved in 50 ml 0.9% saline and 10 ml 2% xylocaine solution then the catheter will be clamped for 6 hours.
  Interventions: Procedure: Group 2 chemical pleurodesis by bleomycin)

INTERVENTIONS:
Procedure: Group 1 (mechanical pleurodesis) — pleural abrasions will be done by scrubbing the parietal and visceral pleura until a uniform aspect of bloody pleura by a piece of gauze attached to the end of a holding forceps , intercostal tube will then placed and monitoring of lung expansion will be done through serial CXR and chest ultrasound follow up and when the lung is fully expanded the tube will be clamped for two hours and follow up CXR will be done for follow up and then the tube removed
  Arms: Group 1 (Mechanical pleurodesis)
Procedure: Group 2 chemical pleurodesis by bleomycin) — Those Patients will have indwelling pleural catheter through which pleural fluid will be drained until dryness and then pleurodesis will be done by 60 mg bleomycin dissolved in 50 ml 0.9% saline and 10 ml 2% xylocaine solution then the catheter will be clamped for 6 hours
  Arms: Group 2 (Chemical pleurodesis by bleomycin)

SUMMARY:
Comparision between pleurodesis by pleural abrasion using medical thoracoscopy and bleomycin instillation via indwelling pleural catheter. Evaluating the effectiveness of pleural abrasion using medical thoracoscopy in patients with malignant pleural effusion and evaluating the role of ROSE in diagnosis and management of malignant pleural effusion

DETAILED DESCRIPTION:
Malignant pleural effusion cause significant morbidity so drainage effusion can provide great palliation and improve quality of life of these patients. There are several diagnostic tools for diagnosing malignant pleural effusion as pleural fluid cytology, closed pleural biopsy or thoracosopic pleural biopsy. Medical thoracoscopy has significant role in diagnosis and management of malignant pleural effusion. Also, pleurodesis may be performed through it by mechanical methods as pleural abrasion or chemical methods by talc poudrage, bleomycin or cisplatin instillation . and surgically through pleurectomy. Recently, using of ROSE (Rapis On-Site Examination) technique during medical thoracoscopy showed high accuracy for distinguishing between benign and malignant lesions, and this help in decision making. In our study, we will use mechanical pleurodesis by pleural abrasion using medical thoracoscpy and chemical pleurodesis by instillation of bleomycin via indwelling pleural catheter.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are 18 years old or more.
* patients with rapidly accumulating moderate & massive malignant pleural. effusion that need frequent aspiration to relieve dyspnea and affect quality of life of the patient.

Exclusion Criteria:

* patients not fit for thoracoscoy.
* patients with life expectency less than 1 month .
* trapped lung (endobronchial lesion).
* excessive pleural adhesios.
* mild effusion not need frequent aspiration and not affect
* quality of life .
* patients with chest infection : pneumonia , empyema .
* patients with performance status that doesn't expected to increase by 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2029-08-10 (Estimated); Study Completion 2029-10-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of successful pleurodesis by chest ultrasound | 6 months
  This will be done every 2 weeks to detect any recollection of fluid in the pleural space. It will be used to determine whether the intervention achieved full or partial success

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed M Abd ElHady, Professor, Study Director — Assiut University Faculty of Medicine
Locations (1):
- Assiut University Faculty of Medicine, Asyut, Egypt

REFERENCES:
- [Background] Bibby AC, Dorn P, Psallidas I, Porcel JM, Janssen J, Froudarakis M, Subotic D, Astoul P, Licht P, Schmid R, Scherpereel A, Rahman NM, Cardillo G, Maskell NA. ERS/EACTS statement on the management of malignant pleural effusions. Eur Respir J. 2018 Jul 27;52(1):1800349. doi: 10.1183/13993003.00349-2018. Print 2018 Jul. PMID 30054348
- [Background] LoCicero J 3rd. Thoracoscopic management of malignant pleural effusion. Ann Thorac Surg. 1993 Sep;56(3):641-3. doi: 10.1016/0003-4975(93)90937-d. PMID 8379759
- [Background] Hamouda D, Elsayed E, Alawady SM. Pleurodesis Using Bleomycin Ampoules, Doxycycline Capsules, and Povidone Iodine Solution in Patients with Malignant Pleural Effusion in Zagazig University Hospitals. 2022;28(5):1022-8.